CLINICAL TRIAL: NCT00515229
Title: Protocol for a Phase II-Study Anti-Inflammatory Pulmonal Therapy of CF-Patients With Amitriptyline and Placebo - Randomised, Double-Blinded, Placebo-Controlled, Cross Over - Study -
Brief Title: Anti-Inflammatory Pulmonal Therapy of CF-Patients With Amitriptyline and Placebo
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: APA-II
Record Dates: First submitted 2007-08-09; First posted 2007-08-13 (Estimated); Last update posted 2007-08-13 (Estimated); Status verified 2007-08

CONDITIONS: Cystic Fibrosis; Infection; Pseudomonas Aeruginosa
Keywords: cystic fibrosis; ceramide; amitriptyline; Pseudomonas aeruginosa; lung function
MeSH Terms: conditions — Cystic Fibrosis; Infections; Pseudomonas Infections | interventions — Amitriptyline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Active Comparator): Verum 1: Each individual capsule has a filling volume of 25 mg amitriptyline, given once an day in the evening over 28 days
  Interventions: Drug: amitriptyline
- 2 (Active Comparator): Verum 1: Each individual capsule has a filling volume of 50 mg amitriptyline, given once an day in the evening over 28 days
  Interventions: Drug: amitriptyline
- 3 (Active Comparator): Verum 3: Each individual capsule has a filling volume of 75 mg amitriptyline, given once an day in the evening over 28 days
  Interventions: Drug: amitriptyline
- 0 (Placebo Comparator): Placebo: Each individual capsule has a filling volume of 25 mg placebo (corn starch), given once an day in the evening over 28 days
  Interventions: Drug: amitriptyline

INTERVENTIONS:
Drug: amitriptyline — Each individual capsule has a filling volume of 25 mg, 50 mg und 75 mg Amitriptyline.
  Placebo: 25 mg corn starch

SUMMARY:
Our data indicate that the CFTR-molecule functions as a transporter for sphingosine-1-phosphate and sphingosine or regulates the uptake of these sphingolipids by epithelial cells. The disturbed uptake of sphingosine and sphingosine-1-phosphate over the cell membrane results in an accumulation of ceramide in the cell membrane, which finally triggers a pro-inflammatory and pro-apoptotic status in the respiratory tract of cystic fibrosis patients. Amitriptyline reduces the cera-mide levels in the lung tissue, normalises the activity of cytokines and prevents constitutive cell death of epithelial cells observed in CFTR-deficient mice. Most important, amitriptyline prevents pulmonary infections of CFTR-deficient mice with P. aeruginosa. These effects of amitriptyline may result in an improved lung function of cystic fibrosis patients.

DETAILED DESCRIPTION:
Cystic fibrosis (CF), the most common autosomal recessive disorder at least in western countries, is caused by mutations of the cystic fibrosis transmembrane conductance regulator molecule (CFTR) and affects approximately 40 000 patients in Europe. Most, if not all, CF-patients develop a chronic pulmonary infection with Pseudomonas aeruginosa (P. aeruginosa). At present it is un-known why CF-patients are highly sensitive to P. aeruginosa infections and, most important, no curative treatment for cystic fibrosis is available.

Our data on CFTR-deficient mice demonstrate that the CFTR-molecule does not only function as a chloride-channel, but also as a transporter for sphingolipids, in particular sphingosine and sphingosine-1-phosphate. Deficiency of functional CFTR in CFTR-knock-out mice results in an alteration of the sphingolipid metabolism in pulmonary epithelial cells and an accumulation of cellular ceramide in these cells.

Inhibition of ceramide release in the lung was achieved by pharmacological and genetic inhibition of the acid sphingomyelinase (ASM) that generates ceramide from sphingomyelin. Amitriptyline was employed to pharmacologically block the ASM genetic inhibition of the ASM was achieved by crossing CFTR- and ASM-deficient mice. Although the ASM is not affected in cystic fibrosis, an inhibition of the enzyme should block the formation of ceramide and, thus, normalize the increase of pulmonary ceramide caused by CFTR-deficiency.

ELIGIBILITY:
Inclusion Criteria:

1. Cystic Fibrosis is proved
2. The patient are older than 18 years (<50 years)
3. No sec discrimination
4. The patient is pulmonal colonized with bacteria
5. Signs of pulmonary exacerbation are not present
6. A full course of therapy is possible without any restrictions
7. Lung function measurement is possible

Exclusion Criteria:

1. Poor metabolizer for amitriptyline (CYP2D6 genotyping)
2. Glaucoma, seizures, heart insufficiency or depression is present
3. Signs of acute pulmonary illness (bronchial or tracheal stenosis, tuberculosis, thorax trauma, acute pneumonia, pneumothorax, bronchial haemorrhage, ARDS) are present
4. intravenous antibiotic treatment was necessary in the last 4 weeks
5. Involvement of the patient in another study
6. Pregnancy

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2006-10; Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Increase in lung function, especially the FEV1 increase | 5 months

SECONDARY OUTCOMES:
Increase of CO-Diffusion | 5 months
Pulmonary Ceramide expression | 5 months
Decrease of cytokine-concentrations | 5 months
Decrease of leukocytes (sputum) | 5 months
Decrease of Pseudomonas | 5 months
Infection parameters in serum | 5 months
Exacerbations | 5 months

CONTACTS AND LOCATIONS:
Overall Officials: Joachim Reithmueller, Dr., Principal Investigator — University of Tuebingen, Paediatric Department
Locations (1):
- University of Tuebingen, Tübingen, Baden-Wurttemberg, Germany

REFERENCES:
- [Derived] Becker KA, Riethmuller J, Luth A, Doring G, Kleuser B, Gulbins E. Acid sphingomyelinase inhibitors normalize pulmonary ceramide and inflammation in cystic fibrosis. Am J Respir Cell Mol Biol. 2010 Jun;42(6):716-24. doi: 10.1165/rcmb.2009-0174OC. Epub 2009 Jul 27. PMID 19635928